CLINICAL TRIAL: NCT05725239
Title: Synchronized Cervical or Auricular VNS With Prefrontal rTMS for Treatment Resistant Depression (TRD)
Brief Title: taVNS or TMS or Both for Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Mark George, Principal Investigator, Medical University of South Carolina
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 00125468
Record Dates: First submitted 2023-01-18; First posted 2023-02-13 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Vagus Nerve Stimulation; Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Vagus Nerve Stimulation (VNS) only (Experimental)
  Interventions: Device: Vagus Nerve Stimulation
- Transcranial Magnetic Stimulation (TMS) only (Experimental)
  Interventions: Device: Transcranial Magnetic Stimulation
- Synchronized VNS and TMS (Experimental)
  Interventions: Device: Vagus Nerve Stimulation; Device: Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Vagus Nerve Stimulation — All taVNS sessions will use the following parameters: 25Hz, 500us pulse width, on for 7 seconds, off for 12 seconds.The length of VNS treatment sessions will be identical to TMS treatment sessions and will have the same 30 minute break between each treatment session. These treatments (active or sham) will be administered to participants each treatment day, for a total of 6 different treatment days, but only 4 are active.
  Arms: Synchronized VNS and TMS; Vagus Nerve Stimulation (VNS) only
Device: Transcranial Magnetic Stimulation — Participants will receive 20 trains of 30 pulses each for a total of 600 pulses per session. We will repeat this for 6 sessions each day, with at least 30 minutes between each session. These treatments (active or sham) will be administered to participants each treatment day, for a total of 6 different treatment days, but only 4 are active, so participants will get 24 TMS sessions over the course.
  Arms: Synchronized VNS and TMS; Transcranial Magnetic Stimulation (TMS) only

SUMMARY:
The purpose of the research is to test out a combined treatment for depression where the investigators stimulate a nerve in the ear while at the same time stimulate the brain with magnets. These treatments are called transcutaneous (through the skin) auricular (ear) vagus nerve stimulation (taVNS) and transcranial (through the skull) magnetic stimulation (TMS). For participants who already have a cervical VNS device, the investigators will not change their treatment and will use this in place of the taVNS. The investigators think this combined method might treat depressive symptoms better than either alone. This study is in person at the Institute of Psychiatry in downtown Charleston on the MUSC campus. First, participants will have a screening session and then will have 6 treatment days total where participants will receive either VNS treatment alone, TMS treatment alone, or both at the same time. The treatment that participants start with will be randomized, and they will have 2 treatment days of each combination.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years old
* Undergoing cervical VNS or have tried and failed two antidepressant medications in the current episode
* Able to provide informed consent
* English speaking and can read and write
* 17-item Hamilton Depression Rating Scale (HAM-D) score ≥20
* Not responding to talking therapy.

Exclusion Criteria:

* Preexisting neurological disorders, or dementia
* History of major head trauma
* Life expectancy <1 year
* Any type of cognitive impairment that would require approval/signature of a legal guardian/representative for participation
* A score of >2 on question 3 of the Hamilton Depression Rating pertaining to suicidality
* Current active suicidal intent or plan, prior attempt within the last 6 months, or who in the judgment of the investigator would be at elevated risk for suicide will be excluded
* Patients who are pregnant will also be excluded. We will require a pregnancy test for individuals of child-bearing potential.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-03-14 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in Hamilton Depression Rating Scale | Through study completion, an average of 8 weeks
  The Hamilton Depression Rating Scale (HDRS) is a commonly used clinician-administered depression rating scale to assess severity of depressive symptoms. The HDRS has a possible score range of 0-52. The higher the HDRS score, the more severe the depressive symptoms are in that patient.
Change in Patient Health Questionnaire 9 | Through study completion, an average of 8 weeks
  The Patient Health Questionnaire 9 (PHQ-9) is a brief self-administered questionnaire to assess depressive symptoms. The PHQ-9 has a possible score range of 0-27. The higher the PHQ-9 score, the more severe the depressive symptoms are in that patient.

SECONDARY OUTCOMES:
Number of adverse outcomes | One week following conclusion of the trial
  Participants will be called at the 1 week and 1 month timepoints following their completion of the trial to inquire about any adverse outcomes they have experienced, if any, since the conclusion of the trial as a means of measuring feasibility of the treatment.
Number of adverse outcomes | One month following conclusion of the trial
  Participants will be called at the 1 week and 1 month timepoints following their completion of the trial to inquire about any adverse outcomes they have experienced, if any, since the conclusion of the trial as a means of measuring feasibility of the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Mark George, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina Institute of Psychiatry, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No